CLINICAL TRIAL: NCT06789510
Title: Treatment of Peyronie's Disease With Platelet-Rich Plasma: A Pilot Study
Brief Title: Treatment of Peyronie's Disease With Platelet-Rich Plasma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Mikael Heering, Medical Doctor, Clinical Assistant, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-24019622-pilot
Record Dates: First submitted 2025-01-15; First posted 2025-01-23 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Peyronies Disease
Keywords: PRP; Platelet-Rich Plasma
MeSH Terms: conditions — Penile Induration | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Each participant will receive six injections (three Platelet-Rich Plasma (PRP) and three saline), administered weekly in a randomized sequence. The RedCap randomization module ("Research Electronic Data Capture", a data management system used for research data) will ensure that each participant receives three injections of each type.
Who Masked: Participant, Investigator
Masking Description: The participant and the investigator/treating doctor will be masked. The syringes will be covered. Only the care provider who prepare the PRP will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet Rich Plasma (PRP) (Experimental): Each participant will receive 3 PRP injections over the 6-week period, with weekly injections in a randomized sequence. The RedCap randomization module will ensure that each participant receives 3 injections of each type.
  Interventions: Other: Autologous Platelet Rich Plasma
- Saline Solution (Placebo) (Placebo Comparator): Each participant will receive 3 saline injections over the 6-week period, with weekly injections in a randomized sequence. The RedCap randomization module will ensure that each participant receives 3 injections of each type.
  In addition, Platelet-Rich Plasma (PRP) will be prepared but, instead of being injected, it will be analyzed for platelet count.
  Interventions: Other: Saline solution

INTERVENTIONS:
Other: Autologous Platelet Rich Plasma — 10 mL PRP intralesional injections will be administered. After the injections, participants will be instructed to perform penile stretching exercises daily until the next injection and to continue these exercises after the final injection until the 3-month follow-up.
  Other Names: PRP
  Arms: Platelet Rich Plasma (PRP)
Other: Saline solution — 10 mL saline solution intralesional injections will be administered. After the injections, participants will be instructed to perform penile stretching exercises daily until the next injection and to continue these exercises after the final injection until the 3-month follow-up.
  Other Names: Placebo
  Arms: Saline Solution (Placebo)

SUMMARY:
The purpose of this pilot study is to optimize a planned randomized, double-blind, placebo-controlled clinical trial evaluating the effects of Platelet-Rich Plasma (PRP) intralesional injections in men affected by Peyronie's disease (PD) in the fibrotic phase. The pilot study aims to identify potential challenges in the practical execution of the clinical trial, particularly regarding PRP preparation and the blinding process. Furthermore, it seeks to evaluate the effects of PRP injections.

DETAILED DESCRIPTION:
The study protocol is structured such that participants, after being informed about the project and providing consent, will attend a baseline visit where relevant data will be collected from the participant, questionnaires, the patient's medical record, and through an objective examination. Subsequently, participants will attend weekly injection sessions for 6 weeks, during which they will receive 3 PRP injections and 3 saline injections (placebo) in a randomized order. Three months after the final injection, participants will attend a follow-up visit, where the final data will be collected. Analysis will then be conducted.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Be able to provide written informed consent
* Diagnosis of PD without active pain and without progressive curvature over the past 3 months (fibrotic phase).
* Penile curvature of 30-95 degrees

Exclusion Criteria:

* Erectile Dysfunction unresponsive to on-demand PDE5 inhibitors
* Hourglass malformation
* Severely calcified plaques where injection is considered unfeasible
* History of priapism.
* History of penile fracture.
* Previous treatment for PD with injections and/or surgery.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Platelet Concentration in the PRP | The 6 week intervention period.
  In the placebo sessions, the Platelet-Rich Plasma (PRP) sample (prepared using the Magellan Autologous Platelet Separator) will be sent for analysis of platelet concentration levels to ensure the quality of the PRP.
Evaluation of the Blinding Process | The 6 week intervention period.
  After each injection, both the administering physician and the participant will be asked to state whether they believe the injection contained PRP or saline. They will also be asked to justify their response, which will allow for adjustments to the practical implementation of the blinding process in the Randomized Controlled Trial (RCT), if necessary.

SECONDARY OUTCOMES:
Adverse Events | From the first injection to the 3 months post intervention follow-up.
  Recording of adverse events following injections to ensure safety. In other studies and clinical practice, no serious adverse events have been reported. However, mild adverse events may include slight pain, ecchymosis, and hematoma.
Degree Changes in Penile Curvature. | From enrollment to 3 months post intervention.
  Dominant curvature angles will be measured using a goniometer based on images of the participants' erect penis (in two planes) at baseline and at follow-up three months after the final injection. The images will be captured in the outpatient clinic following the administration of Alprostadil to ensure high quality and consistency.
Changes in Plaque Size | From enrollment to 3 months post intervention.
  Plaque size will be measured at baseline and three months after the final injection using a ruler, calculated as the product of plaque length and width. Participants with more than two plaques or with significant plaque heterogeneity will not have plaque size measured and will be excluded from these analyses but may still participate in the study.
Changes in the Peyronie's Disease Questionnaire (PDQ) | From enrollment to 3 months post intervention.
  The Peyronie's Disease Questionnaire (PDQ) is a 15-question self-reported survey that measures the impact and severity of Peyronie's disease (PD) symptoms in 3 domains, including psychological and physical symptoms, penile pain and symptom bother.
  Higher domain scores indicate a greater negative impact. The range of scores for each domain is 0 to 24 for PD psychological and physical symptoms, 0 to 30 for penile pain and 0 to 16 for PD symptom bother.
  The participants will complete the survey at baseline and three months after the final injection.
Changes in the Erection Hardness Score (EHS) | From enrollment to 3 months post intervention.
  The participants will rate the hardness of their erection via the single-item Likert scale EHS, at baseline and three months after the final injection. The scale is from 0-4. 0 is no erection, the higher the score the better erection.
Changes in the Major Depression Inventory (MDI) | From enrollment to 3 months post intervention.
  The Major Depression Inventory (MDI) is a patient-reported outcome measure to assist with diagnosing and evaluation of the severity of a patient's depression.
  The MDI score ranges from 0 to 50, where 0 represents no depression symptoms and 50 represents the most severe depression symptoms.
  The participants will complete the MDI questionnaire at baseline and three months after the final injection.
  The MDI is included due to previously described associations between Peyronie's disease and depression. The data may be used to assess the impact of disease progression on potential depressive symptoms.
The Ability to Engage in Sexual Intercourse (question) | From enrollment to 3 months post intervention.
  The participants will be assessed at baseline and three months after the final injection regarding their ability to engage in sexual intercourse. This will be assessed by asking participants a single binary question: whether they are able to engage in sexual intercourse (yes or no).
Preference for Surgical Intervention (question) | From enrollment to 3 months post intervention.
  The participants will be inquired about their preference for surgical intervention in relation to the current penile curvature at baseline and 3 months after the final injection. This will be assessed by asking participants a single binary question: whether they wish to undergo surgery given their current curvature (yes or no).
Satisfaction | From enrollment to 3 months post intervention.
  The participants will complete a Global Assessment Scale Questionnaire regarding overall treatment satisfaction at the 3-month follow-up after the final injection.
  The questionnaire consists of a single question regarding the participants' overall satisfaction with the treatment, to be answered on a scale from 1 to 5. A higher value indicates greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev and Gentofte University Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No